CLINICAL TRIAL: NCT01093937
Title: A 10-Week Pilot Study of Varenicline (Champix) Versus Placebo for Smoking Cessation/Reduction in Patients With Bipolar Disorder
Brief Title: Study of Varenicline (Champix) for Smoking Cessation/Reduction in Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Tobacco Control Research Initiative (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Tony P. George, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 229/2009
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Nicotine Dependence
Keywords: Bipolar disorder; Bipolar-I; Varenicline; Champix; Chantix; Nicotine; Nicotinic receptor; Nicotinic receptor dysregulation; Dopamine; Acetylcholine; Cigarette; Smoking; Tobacco; Dependence; Neuropsychological function
MeSH Terms: conditions — Tobacco Use Disorder; Bipolar Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: varenicline — One to four 0.5 mg capsules (0.5-2.0 mg) orally per day for ten weeks.
  Other Names: Champix; Chantix

SUMMARY:
Bipolar Disorder is a chronic relapsing mental disorder characterized by periods of elevated, expansive and irritable mood, often alternating with periods of significant clinical depression. People with Bipolar Disorder are typically heavy smokers who have difficulty quitting, and this is associated with significant tobacco-related medical illness and death.

The proposed study will be a double-blind, placebo-controlled 10-week clinical trial of the safety and efficacy of varenicline (Champix™) in thirty subjects with Bipolar I Disorder. This medication is the latest first-line pharmacotherapy for smoking cessation and has been shown to be efficacious for smoking cessation, but has not yet been systematically studied in persons with Bipolar Disorder.

DETAILED DESCRIPTION:
Varenicline (VAR) is a α4β2 central nicotinic acetylcholine receptor (nAChR) partial agonist. It is believed to mimic the effect of nicotine by stimulating nAChRs and releasing sufficient dopamine in order to reduce craving and withdrawal effects. In the past two years since the approval of VAR there have been some increasing concerns about this medication, particularly in psychiatric smokers. Besides the typical side effects of nausea and insomnia, it has been associated with treatment-emergent suicidality, aggression, psychosis, and induction of hypomania or mania.

Study Design:

Thirty nicotine-dependent cigarette smokers with Bipolar I Disorder will be enrolled (N=30). All subjects will be symptomatically stable prior to enrollment, and compliant with their mood-stabilizer medication treatment to minimize the chances of adverse outcomes. The treatment group would receive flexible doses of varenicline (VAR) ranging from one to four capsules (0.5-2.0 mg) orally per day. The control group would receive one to four capsules of placebo VAR (0 mg) orally per day. All subjects would receive weekly Cognitive Behavioral Therapy (CBT) offered in group format to help them deal with tobacco cravings and mood management. The target quit date would be set during Week 3 of the trial. Comprehensive neuropsychological assessment and laboratory testing will be given at baseline and ten weeks;

Hypotheses:

1. Varenicline will be superior to placebo for smoking cessation outcomes.
2. Varenicline will be well-tolerated and safe for use in Bipolar I smokers in comparison to placebo.
3. Varenicline will reduce smoking indices (Carbon monoxide, cotinine) and have minimal effects on psychiatric symptomatology in mood-stabilizer treated Bipolar I smoking patients.
4. The presence of prefrontal cortical, impulsivity and attentional deficits on the baseline neuropsychological battery will predict smoking cessation treatment failure in Bipolar I smokers.

Significance:

* This would be the first placebo-controlled clinical trial using varenicline for the treatment of tobacco dependence in people with Bipolar Disorder.
* There is an immense need for a safe and effective smoking cessation therapy for smokers with bipolar illness. The co-morbidity between the major psychiatric disorders and nicotine dependence has been well established. The prevalence of cigarette smoking in patients with bipolar disorder is approximately 50-70% as compared to ~19% in the Canadian population. Moreover, smokers with Bipolar Disorder suffer to a higher extent from smoking-related illnesses than non-psychiatric smokers.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview (SCID) derived DSM-IV diagnoses of Bipolar Disorder (Type I or II), and Nicotine Dependence
* Young Mania Rating Scale Total Score <12 at study entry
* HAM-D 17-Item Score >5 and <24 at study entry
* Fagerstrom Test for Nicotine Dependence (FTND) score of 5 or higher
* Be able to provide informed consent to participate in this study as judged by clinical evaluation, and scoring at least 80% on a post-consent "test"
* Smoking at least 10 cigarettes per day (confirmed by an expired breath CO level >10 ppm and a plasma cotinine level >150 ng/ml at baseline)
* Be motivated to quit smoking within 30 days of initial evaluation, as assessed by a score of 7 or higher on the Contemplation Ladder assessment tool
* On a stable dose of a mood stabilizer for at least 1 month (e.g. lithium, valproate, carbamazepine, atypical antipsychotic)
* Judged by the study psychiatrists and/or trained psychiatric clinicians to be in remission from active manic, hypomanic, major depressive and psychotic symptoms based on a clinical interview and SCID-IV ≥1 month prior to study enrollment

Exclusion Criteria:

* Meet criteria for current abuse or dependence for any other alcohol or illicit substance within the past 3 months of study enrollment
* Current evidence by SCID-IV and clinical evaluation of suicidality, homicidality or psychosis
* Meet DSM-IV criteria for current major depression at the time of baseline evaluation
* A history of hypersensitivity or other known adverse reactions (e.g. hyperstimulation, severe agitation) to varenicline.
* Serious medical conditions (i.e. a history of severe cardiac, renal or hepatic disease, diabetes mellitus or thyroid abnormalities)
* EKG abnormalities
* Prescription of Nicotine Replacement Therapies (NRTs) including patches, gum, lozenges or inhalers
* Prescription of monoamine oxidase inhibitors (MAO-I's) including selegiline or moclobemide
* Prescription of varenicline
* Prescription of bupropion SR
* The presence of manic, mixed manic or hypomanic symptoms in the past one month prior to study enrollment.
* A lifetime history of antidepressant-induced mania or hypomania
* A history of suicidal ideation while taking antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety | Baseline (week 0), Weeks 1-9, End of trial (Week 10)
  Medical and psychiatric evaluation
Smoking cessation | End of trial (Week 10)
  Medical and psychiatric evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research